CLINICAL TRIAL: NCT03422627
Title: A Phase 1b/2 Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Efavaleukin Alfa in Adult Subjects With Steroid Refractory Chronic Graft Versus Host Disease
Brief Title: Safety and Efficacy of Efavaleukin Alfa in Subjects With Steroid Refractory Chronic Graft Versus Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160283; 2017-000763-33 (EudraCT Number)
Record Dates: First submitted 2018-01-16; First posted 2018-02-06 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Chronic Graft Versus Host Disease cGVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Efavaleukin Alfa Multiple Ascending Doses (Experimental): Efavaleukin will be administered as multiple ascending doses (MAD) across cohorts 1-5. Each dosing cohort will consist of between 3 and 6 subjects who will receive efavaleukin alfa subcutaneously (SC) either every week or every 2 weeks plus protocol permitted background therapy for 52 weeks. At the discretion of the Sponsor, following discussion and agreement between the principal investigator and medical monitor, subjects responding to efavaleukin alfa (as assessed by the end of week 50), who wish to continue treatment, may continue to receive efavaleukin alfa treatment at their current dosing regimen.
  Interventions: Drug: Efavaleukin Alfa
- Phase 2: RP2D Efavaleukin Alfa (Experimental): The phase 2 portion of this study will be conducted as a single arm, multi-center, open label trial in subjects with steroid refractory chronic graft versus Host Disease (cGVHD). All subjects will receive the recommended phase 2 dose (RP2D) of efavaleukin alfa for up to 52 weeks plus protocol permitted background therapy for cGVHD.
  Due to early study termination the Phase 2 portion of the study was never opened.
  Interventions: Drug: Efavaleukin Alfa

INTERVENTIONS:
Drug: Efavaleukin Alfa — Phase 1: This study will be conducted as a multiple ascending dose (MAD) study. Each dosing cohort will consist of between 3 and 6 subjects who will receive efavaleukin alfa subcutaneously (SC) either every week or every 2 weeks plus protocol permitted background therapy for 52 weeks. At the discretion of the Sponsor, following discussion and agreement between the principal investigator and medical monitor, subjects responding to efavaleukin alfa (as assessed by the end of week 50), who wish to continue treatment, may continue to receive efavaleukin alfa treatment at their current dosing regimen for up to an additional 208 weeks through an extended dosing period. All subjects who continue to receive efavaleukin alfa during the extended dosing period will be reevaluated every 6 months for their response to treatment.
  Phase 2: All subjects will receive the recommended phase 2 dose (RP2D) of efavaleukin alfa for 52 weeks.
  Other Names: AMG 592

SUMMARY:
Phase 1b: To evaluate the safety and tolerability of multiple ascending doses of efavaleukin alfa in subjects with steroid refractory chronic graft versus host disease (cGVHD).

Phase 2: To evaluate the efficacy of efavaleukin alfa in subjects with steroid refractory cGVHD as measured by overall response rate (ORR) at 16 weeks according to the 2014 cGVHD NIH Consensus Criteria.

Due to early termination, the Phase 2 portion of this study was not conducted.

ELIGIBILITY:
Inclusion Criteria Subjects are eligible to be included in the study only if all of the following criteria apply:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Subject is an adult ≥ 18 years old at the time of signing the informed consent.
* Subject is a recipient of an allogeneic HSCT.
* Subject has moderate to severe steroid-refractory cGVHD as defined by all of the following criteria:
* Diagnosed with cGVHD per the 2014 cGVHD NIH Consensus Criteria
* Steroid refractory cGVHD, defined as having persistent signs and symptoms of cGVHD despite ≥ 4 weeks of prednisone (or equivalent) dosed at ≥ 0.25 mg/kg/day (or ≥ 0.5 mg/kg every other day).
* Moderate to severe cGVHD (in accordance with 2014 cGVHD NIH Consensus Criteria at screening with involvement of at least one of the following organs at the screening and baseline visits: skin, mouth, eyes, gastrointestinal (GI) tract, liver, lungs, and joint and fascia.
* Subject has received no more than 3 previous treatments for cGVHD, excluding topical agents.
* Treatment with corticosteroids is considered a treatment for cGVHD and should be included in determining the number of previous treatments.
* Lines of therapy consisting of concurrent medications or interventions (eg, tacrolimus and corticosteroids; ECP and corticosteroids) count as 2 separate treatments.
* If cGVHD has worsened during a taper of immunosuppressive agents, restoring the agents to therapeutic level is permitted and does not count as an additional treatment.
* Subject may be receiving corticosteroid therapy provided that the dose is ≤ 1 mg/kg/day of systemic prednisone or equivalent and has been stable for at least 2 weeks prior to first dose of efavaleukin alfa.
* Subject may be receiving other non-corticosteroid immunosuppressive therapies provided that the immunosuppressant dose is stable for at least 2 weeks prior to first dose of efavaleukin alfa. Adjustments to dose of calcineurin inhibitor or sirolimus are allowed only to maintain drug levels within therapeutic range.
* Subject has a Karnofsky performance status score ≥ 50%.
* Subject has an estimated life expectancy of > 3 months.
* Subject must have adequate hepatic function, defined below, unless the treating physician documents the abnormal LFTs as consistent with hepatic cGVHD:
* total bilirubin < 2.0 mg/dL (34.2 mol/L) [elevated values due to Gilbert's Syndrome or of non- hepatic origin are excluded].
* aspartate transaminase [AST; SGOT]/Alanine transaminase [ALT; SGPT] ≤ 2x upper limit of normal (ULN).
* If LFT abnormalities are deemed consistent with hepatic cGVHD by the investigator, a liver biopsy will not be mandated.
* Subject must have adequate pulmonary function defined as: forced expiratory volume in 1 second (FEV1) ≥ 50% or hemoglobin-adjusted diffusion capacity for carbon monoxide (DLCO Hb) ≥ 40% of predicted, unless pulmonary dysfunction is deemed to be due to cGVHD.
* Subject must have adequate renal function defined as: a calculated glomerular filtration rate of > 50 mL/min/1.73 m2 using the MDRD formula.
* Subject must have adequate cardiac function defined as: no history within 6 months prior to screening of myocardial infarction, unstable angina, New York Heart Associate Class III or IV heart failure, or stroke. No findings on the screening electrocardiogram (ECG) that in the opinion of the investigator requires further cardiovascular evaluation, including severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Subject must have adequate bone marrow function indicated by ANC > 1.00 x 109/L and platelets > 50 x 109/L without growth factors or transfusions within the 4 weeks prior to starting efavaleukin alfa.

Exclusion Criteria Subjects are excluded from the study if any of the following criteria apply.

* Subject is concurrently receiving treatment with calcineurin-inhibitor plus sirolimus (either agent alone is acceptable).
* Subject has received ibrutinib, imatinib, bortezomib, entospletinib, ruxolitinib or other JAK inhibitor, or treatment with any investigational drug or device within 4 weeks prior to starting efavaleukin alfa.
* Subject has received treatment with T-cell depleting, B-cell depleting or IL-2 signaling targeted medication (eg, ATG, alemtuzumab, basiliximab, denileukin diftitox, IL-2, rituximab) within 12 weeks prior to starting efavaleukin alfa.
* Subject has received treatment with T regulatory cell expanding therapies (ie PUVA, UVB, adoptively transferred T regulatory cells) within 4 weeks prior to starting efavaleukin alfa.
* Subject has received a donor lymphocyte infusion within 12 weeks prior to starting dose of efavaleukin alfa.
* Subject with active morphologic relapse/progression of hematologic malignancy post transplantation. Persistent CLL early after transplantation that subsequently entered remission will not be excluded.
* Subject has a history of malignancy, other than the indication for hematopoietic cell transplantation, with the following exceptions:
* adequately treated nonmelanoma skin cancers without current evidence of disease
* adequately treated cervical carcinoma in situ without current evidence of disease
* adequately treated breast ductal cancer in situ without current evidence of disease
* any malignancy treated with curative intent and with no evidence of active disease present for more than 5 years prior to screening and felt to be at low risk for recurrence by the treating physician
* Subject has a history of thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura.
* Subject has an active infection requiring treatment with IV antibiotics or has been hospitalized for treatment of an active infection in the 4 weeks prior to starting dose of efavaleukin alfa.
* Subject has known history of active tuberculosis.
* Positive test for tuberculosis during screening defined as either:
* positive purified derivative (PPD) (≥ 5 mm of induration at 48 to 72 hours after test is placed) OR
* positive Quantiferon or T-SPOT test o a positive PPD and a history of Bacillus Calmette-Guérin vaccination are allowed with a negative Quantiferon or T-SPOT test and negative chest x-ray

  * a positive PPD test (without a history of Bacillus Calmette-Guérin vaccination) or a positive

Quantiferon or T-SPOT test are allowed if they have ALL of the following at screening:

* no symptoms per tuberculosis worksheet provided by Amgen
* document history of a completed course of adequate prophylaxis (completed treatment for latent tuberculosis per local standard of care prior to the start of investigational product
* no known exposure to a case of active tuberculosis after most recent prophylaxis
* negative chest X-ray o an indeterminate Quantiferon or T-SPOT test is allowed if they have ALL of the following at screening:
* no symptoms per tuberculosis worksheet provided by Amgen
* no known recent exposure to a case of active tuberculosis
* no history of a positive Quantiferon or T-SPOT test without documented history of a completed course of adequate prophylaxis (completed treatment for latent tuberculosis per local standard of care prior to the start of investigational product)
* negative chest X-ray
* are deemed to be at low risk for tuberculosis exposure in the opinion of the principle investigator
* Subject is positive for hepatitis B surface antigen, hepatitis B core antibody (confirmed by hepatitis B deoxyribonucleic acid [DNA] polymerase chain reaction [PCR] test) or detectable hepatitis C virus ribonucleic acid (RNA) by PCR (screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive). Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed.
* Subject has positive test results for Human Immunodeficiency Virus (HIV) or known to be HIV-positive.
* Phase 1b subject has a drug or alcohol urine test positive for illicit drugs at the screening visit. Prescription medications detected by the drug test are allowed if they are being taken under the direction of a physician or if permitted for recreational purposes as per country regulations..
* Phase 1b subject cannot be a current smoker, nor have used any nicotine or tobacco containing products within the last 6 months prior to screening. These types of products include but are not limited to: snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches.
* Phase 1b subject is unable to avoid alcohol during the 4-week DLT evaluation period or tobacco consumption for the duration of the study.
* Subject has known sensitivity to efavaleukin alfa or its excipients to be administered during dosing.
* Subject likely to be unable to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments [COAs]) to the best of the subject and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Females who are pregnant or breastfeeding, or planning to become pregnant or breastfeed during treatment and for an additional 6 weeks after the last dose of efavaleukin alfa.
* Females of child-bearing potential with a positive pregnancy test (assessed by a serum pregnancy test at screening and a urine pregnancy test at baseline).
* Females of childbearing potential who are unwilling to use 1 highly effective method of contraception during treatment and for an additional 6 weeks after receiving the last dose of efavaleukin alfa.
* Subject has previously entered the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Ohio State University Wexner Medical Center Arthur G James Cancer Hospital and Solove Research, Columbus, Ohio
  - Texas Oncology Baylor, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Belgium
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Saint Louis, Paris
- Japan (3):
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into this study at sites in Belgium, France, Japan, and the United States.
Pre-assignment Details: Screening tests and procedures were performed up to 28 days preceding treatment. The study was planned to have a Phase 1b part and a Phase 2 part. The study was cancelled before enrolling participants into the Phase 2 part. Therefore, results presented only include data for the Phase 1b part.
Groups:
- Cohort 1: Participants in Cohort 1 received efavaleukin alfa subcutaneously (SC) once every 2 weeks (Q2W) plus protocol permitted background therapy for 52 weeks. Four ascending dose levels of efavaleukin alfa were administered between the 5 cohorts as follows. Dose 1 (low dose), dose 2 (low-mid dose), dose 3 (high-mid dose), dose 4 (high dose). Participants in Cohort 1 received dose 2.
  At the discretion of the sponsor, following discussion and agreement between the principal investigator and medical monitor, participants that responded to efavaleukin alfa were permitted to continue to receive efavaleukin alfa treatment at their current dosing regimen for up to a maximum of 258 weeks (Q2W dose), if they remained eligible for extended dosing. Participants then completed the 6-week safety follow up after their last dose of efavaleukin alfa.
- Cohort 2: Participants in Cohort 2 received efavaleukin alfa SC once every week (QW) plus protocol permitted background therapy for 52 weeks. Four ascending dose levels of efavaleukin alfa were administered between the 5 cohorts as follows. Dose 1 (low dose), dose 2 (low-mid dose), dose 3 (high-mid dose), dose 4 (high dose). Participants in Cohort 2 received dose 1.
  At the discretion of the sponsor, following discussion and agreement between the principal investigator and medical monitor, participants that responded to efavaleukin alfa were permitted to continue to receive efavaleukin alfa treatment at their current dosing regimen for up to a maximum of 259 weeks (QW dose), if they remained eligible for extended dosing. Participants then completed the 6-week safety follow up after their last dose of efavaleukin alfa.
- Cohort 3: Participants in Cohort 3 received efavaleukin alfa SC Q2W plus protocol permitted background therapy for 52 weeks. Four ascending dose levels of efavaleukin alfa were administered between the 5 cohorts as follows. Dose 1 (low dose), dose 2 (low-mid dose), dose 3 (high-mid dose), dose 4 (high dose). Participants in Cohort 3 received dose 3.
  At the discretion of the sponsor, following discussion and agreement between the principal investigator and medical monitor, participants that responded to efavaleukin alfa were permitted to continue to receive efavaleukin alfa treatment at their current dosing regimen for up to a maximum of 258 weeks (Q2W dose), if they remained eligible for extended dosing. Participants then completed the 6-week safety follow up after their last dose of efavaleukin alfa.
- Cohort 4: Participants in Cohort 4 received efavaleukin alfa SC QW plus protocol permitted background therapy for 52 weeks. Four ascending dose levels of efavaleukin alfa were administered between the 5 cohorts as follows. Dose 1 (low dose), dose 2 (low-mid dose), dose 3 (high-mid dose), dose 4 (high dose). Participants in Cohort 4 received dose 2.
  At the discretion of the sponsor, following discussion and agreement between the principal investigator and medical monitor, participants that responded to efavaleukin alfa were permitted to continue to receive efavaleukin alfa treatment at their current dosing regimen for up to a maximum of 259 weeks (QW dose), if they remained eligible for extended dosing. Participants then completed the 6-week safety follow up after their last dose of efavaleukin alfa.
- Cohort 5: Participants in Cohort 5 received efavaleukin alfa SC Q2W plus protocol permitted background therapy for 52 weeks. Four ascending dose levels of efavaleukin alfa were administered between the 5 cohorts as follows. Dose 1 (low dose), dose 2 (low-mid dose), dose 3 (high-mid dose), dose 4 (high dose). Participants in Cohort 5 received dose 4.
  At the discretion of the sponsor, following discussion and agreement between the principal investigator and medical monitor, participants that responded to efavaleukin alfa were permitted to continue to receive efavaleukin alfa treatment at their current dosing regimen for up to a maximum of 258 weeks (Q2W dose), if they remained eligible for extended dosing. Participants then completed the 6-week safety follow up after their last dose of efavaleukin alfa.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 7 | 7 | 7 | 6 | 5
Completed up to Week 52 and Opted for Extended Dosing | 2 | 1 | 2 | 3 | 0
Completed up to Week 52 and Did Not Opt for Extended Dosing | 0 | 1 | 1 | 0 | 1
Completed | 2 | 2 | 3 | 3 | 1
Not Completed | 5 | 5 | 4 | 3 | 4
Not completed — Protocol-specified Criteria | 1 | 1 | 0 | 0 | 2
Not completed — Requirement for Alternative Therapy | 1 | 1 | 2 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 2
Not completed — Ineligibility Determined | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Measured in the safety analysis set, which included all participants who received at least 1 dose of efavaleukin alfa.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 5 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.5) | 52.9 (17.4) | 49.4 (12.2) | 55.3 (7.6) | 64.6 (5.9) | 53.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 1 | 12
  Male | 4 | 4 | 5 | 3 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 5 | 6 | 6 | 5 | 23
  Unknown or Not Reported | 5 | 2 | 1 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 4 | 4 | 4 | 3 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 1 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: A DLT was defined as a:
  * Non-hematological toxicity ≥grade-4(per common terminology criteria for adverse events [CTCAE] v4.03) related to efavaleukin alfa. Non-hematological lab abnormalities without clinical significance weren't considered DLTs.
  * Hematological toxicity ≥grade 4 related to efavaleukin alfa defined as decreases in peripheral counts (absolute neutrophil count or platelets) persisting longer than 72 hrs, as measured by 2 separate results, that were not related to malignant disease relapse, infection, or other etiologies.
  * Constitutional events (ie, fever, fatigue) ≥grade 3 that were classified as serious adverse events by the investigator and related to efavaleukin alfa.
  * Infection is considered an expected complication of chronic graft versus host disease (cGVHD) and its treatment. Only grade 4 or 5 infections considered by the investigator to be related to efavaleukin alfa were reviewed by the dose level review meeting to determine whether it was considered a DLT.
Time Frame: Up to 4 weeks after first dose of study drug administration
Population: Measured in the DLT analysis set, which included DLT-evaluable participants in the phase 1b portion of the study. To be evaluable for a DLT participants must have received at least 2 doses of efavaleukin alfa or have experienced a DLT within the DLT evaluation period. The DLT evaluation period was defined as 4 weeks after the first dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Treatment-related Adverse Event (AE)
Description: A treatment-related AE was any untoward medical occurrence in a clinical study participant deemed to have a possibly causal relationship to the study treatment as determined by the investigator.
Time Frame: Day 1 until the end of study; median (min, max) duration was 38.01 (3.27, 139.81) weeks
Population: Measured in the safety analysis set, which included all participants who received at least 1 dose of efavaleukin alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 5
Participants | 5 | 5 | 6 | 6 | 4

3. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Treatment-emergent AE
Description: A treatment-emergent AE was any untoward medical occurrence in a clinical study participant that occurred after first dose.
Time Frame: Day 1 until the end of study; median (min, max) duration was 38.01 (3.27, 139.81) weeks
Population: Measured in the safety analysis set, which included all participants who received at least 1 dose of efavaleukin alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 5
Participants | 6 | 6 | 7 | 6 | 4

4. Primary Outcome: Phase 1b: Number of Participants Who Experienced a Treatment-emergent Serious AE
Description: A treatment-emergent serious AE was any untoward medical occurrence in a clinical study participant that occurred after first dose that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or another medically important serious event.
Time Frame: Day 1 until the end of study; median (min, max) duration was 38.01 (3.27, 139.81) weeks
Population: Measured in the safety analysis set, which included all participants who received at least 1 dose of efavaleukin alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 5
Participants | 5 | 3 | 3 | 4 | 3

ADVERSE EVENTS:
Time Frame: Mortality: from enrollment until the end of study; median (min, max) duration was 38.44 (3.56, 140.09) weeks. Serious and non-serious adverse events: from Day 1 until the end of study; median (min, max) duration was 38.01 (3.27, 139.81) weeks.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/7 | 1/7 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/7 | 3/7 | 3/7 | 4/6 | 3/5
Other Adverse Events (participants affected / at risk) | 6/7 | 6/7 | 7/7 | 6/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=7) | Cohort 3 (N=7) | Cohort 4 (N=6) | Cohort 5 (N=5)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 2
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=7) | Cohort 2 (N=7) | Cohort 3 (N=7) | Cohort 4 (N=6) | Cohort 5 (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Meibomianitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral lichen planus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 0 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 3 | 1 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 2 | 0
Injection site rash (General disorders) | 0 | 1 | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 2 | 4 | 2 | 2
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 1 | 2
Pyrexia (General disorders) | 2 | 1 | 2 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Acute graft versus host disease oral (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 2 | 1 | 0 | 0 | 0
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 1 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Graft versus host disease in eye (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Graft versus host disease in skin (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal disease carrier (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Keratitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pathogen resistance (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Enterovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 1 | 0
Human rhinovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Zinc deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cervix oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pharyngeal enanthema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03422627/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT03422627/SAP_001.pdf